CLINICAL TRIAL: NCT00997009
Title: Randomized Phase II Study of Carboplatin and Paclitaxel +/- Cetuximab, in Advanced and/or Recurrent Cervical Cancer
Brief Title: Study of Adding Cetuximab to Chemotherapy for the Treatment of Advanced and/or Recurrent Cervical Cancer
Acronym: MITO CERV 2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITO CERV 2; 2009-010099-74 (EudraCT Number)
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-03

CONDITIONS: Cervical Cancer
Keywords: EGFR; chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Carboplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): chemotherapy plus cetuximab
  Interventions: Drug: paclitaxel; Drug: carboplatin; Drug: cetuximab
- Arm B (Active Comparator): chemotherapy
  Interventions: Drug: paclitaxel; Drug: carboplatin

INTERVENTIONS:
Drug: paclitaxel — 175 mg/m2 IV day 1, every 21 days
Drug: carboplatin — AUC 5 IV day 1 every 21 days
Drug: cetuximab — 400 mg/m2 IV, one week before starting carboplatin and paclitaxel; then 250 mg/m2 IV day 1, weekly
  Arms: Arm A

SUMMARY:
This study aims to assess the activity of a combination of cetuximab (weekly) with carboplatin + paclitaxel (every three weeks) comparing it to chemotherapy alone in terms of event-free survival (EFS).

DETAILED DESCRIPTION:
The poor long-term results in the standard treatment of chemotherapy for cervical cancer make research into new, more beneficial treatment strategies necessary. Cetuximab is a new type of drug that blocks the epidermal growth factor receptor (anti-EFGR), and has shown significant activity in other cancers (colon, head and neck) where expression of EGFR is high. Cervical cancer cells express EGFR in a very high proportion of cases, especially in recurrent or resistant disease. This study evaluates the activity of the addition of cetuximab to full doses of carboplatin and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Advanced and/or metastatic cervical cancer patients untreated or having failed only one previous chemotherapy (with at least 6 months of progression free interval, with or without concomitant or sequential radiotherapy).
* At baseline, presence of at least one measurable target lesion (a lesion that can be accurately measured in at least one dimension i.e. longest diameter at least 20 mm with conventional CT scan or at least 10 mm with spiral CT scan according to RECIST Criteria).
* Not amenable to surgery and/or radiotherapy.
* PS 0-1 according to ECOG.
* Age >18.
* Life expectancy of at least 3 months.
* Adequate organ functions

  * Hematopoietic: Leukocytes > 3,000/mm3; Absolute neutrophil count > or = 1,500/mm3; Platelets count > or = 100,000/mm3; Hemoglobin > or = 9 g/dL
  * Hepatic: AST and ALT < or = 3 times upper limit of normal (ULN)*; Alkaline phosphatase < or = 3 times ULN*; Bilirubin < or = 1.5 times ULN

    *: < or = 5 times ULN if liver metastases are present
  * Renal: Creatinine clearance > or = 45 mL/min
* No other invasive malignancy within the past 5 years except non-melanoma skin cancer.
* All radiology studies must be performed within 28 days prior to randomization.
* Absence of any psychological, familial, sociological or geographical conditions potentially hampering compliance with the study protocol and follow-up schedule.
* Written informed consent.

Exclusion Criteria:

* Pregnant (potentially fertile patients must use contraceptive measures to avoid pregnancy during and for at least 3 months after study participation and must have a negative serum pregnancy test at baseline).
* Patients should not be breast-feeding during treatment and for 2 months following the end of treatment.
* More than one previous chemotherapy line.
* Active infection requiring antibiotics.
* Symptomatic peripheral neuropathy >grade 2 according to the CTCAE.
* Congestive heart failure or angina pectoris even if it is medically controlled. Previous history of myocardial infarction within 1 year from study entry, uncontrolled high risk hypertension or arrhythmia.
* Known hypersensitivity to the study drugs or to drugs with similar chemical structures.
* Concurrent treatment with other experimental drugs.
* Participation in another clinical trial with any investigational drug within 30 days prior to study screening.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2009-10; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
event free survival | after 3 and 6 cycles of treatment (each cycle is 21 days), and every 3 months thereafter up to 18 months

SECONDARY OUTCOMES:
adverse events | after each treatment cycle (each cycle is 21 days) up to 30days
  according CTCAE criteria
overall survival | 18 months
skin toxicity and correlation with cetuximab activity | after 3 and 6 cycles of therapy (each cycle is 21 days), and every 3 months thereafter up to 18 months
EGFR/KRAS expression and correlation with cetuximab activity | at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Alessandro Morabito, M.D.,, Principal Investigator — National Cancer Institute, Naples; Ciro Gallo, M.D., Ph.D., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (15):
- Italy (15):
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Ospedale Oncologico A. Businco, Cagliari
  - Universita Cattolica del Sacro Cuore, Campobasso
  - Istituto Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Nazionale Tumori, Milan
  - A.O. Unversitaria Policlinico, Modena
  - Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Uro-Ginecologico, Napoli
  - A.O. Universitaria Federico II, Napoli
  - Seconda Università di Napoli, Napoli
  - Istituto Oncologico Veneto, Padua
  - Ospedale Silvestrini, Perugia
  - Istituto Regina Elena, Roma
  - Universita Cattolica del Sacro Cuore, Roma
  - Ospedale S. Chiara, Trento
  - A.O. di Udine S. Maria della Misericordia, Udine